CLINICAL TRIAL: NCT05676853
Title: A Phase 3 Open-Label Study of Safety of Weekly Subcutaneous Pegzilarginase in Subjects With Arginase 1 Deficiency
Brief Title: A Study of Safety of Weekly Subcutaneous Pegzilarginase in Subjects With Arginase 1 Deficiency
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Aeglea Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAEB1102-305
Record Dates: First submitted 2022-12-21; First posted 2023-01-09 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Arginase I Deficiency; Hyperargininemia
Keywords: ARG1-D
MeSH Terms: conditions — Hyperargininemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pegzilarginase (Experimental): Weekly subcutaneous dosing of pegzilarginase plus individualized disease management for 52 weeks
  Interventions: Drug: Pegzilarginase

INTERVENTIONS:
Drug: Pegzilarginase — Individualized disease management which includes severe protein restriction, essential amino acid supplementation and the ammonia scavengers when indicated
  Other Names: Co-ArgI-PEG; AEB1102

SUMMARY:
This is an open-label, multicenter study to evaluate the safety of weekly SC administration of pegzilarginase over 12 months in subjects with ARG1-D. The study consists of a screening period of up to 4 weeks, a subsequent 12-month treatment period, and a Safety Follow-Up Visit 2 weeks after the last treatment.

DETAILED DESCRIPTION:
Open-label, multicenter study to evaluate the safety of weekly SC administration of pegzilarginase over 12 months in subjects with ARG1-D. The study consists of a screening period of up to 4 weeks, a subsequent 12-month treatment period, and a Safety Follow-Up Visit 2 weeks after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Prior enrollment in pegzilarginase clinical studies, with completion of treatment or continued dosing as of the study termination date
2. Written informed consent by subject/parent/legal guardian, which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol
3. Negative pregnancy test within 7 days prior to dosing in childbearing subjects if they are sexually active
4. If the subject (male or female) is engaging in sexual activity that could lead to pregnancy, must be surgically sterile, post-menopausal (female), or must agree to use a highly effective method of birth control during the study and for a minimum of 30 days after the last study drug administration. Highly effective methods of contraception include combined (estrogen and progestogen-containing) hormonal contraception associated with inhibition of ovulation, progesterone-only hormonal contraception associated with inhibition of ovulation, intrauterine device, or intrauterine hormone-releasing system

Exclusion Criteria:

1. Subjects with acute or ongoing hyperammonemia within 6 weeks of the first dose
2. Subjects with medical conditions or underlying issues that, in the opinion of the Investigator, would preclude participation in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events | Baseline through week 54
  To evaluate the safety of long-term subcutaneous pegzilarginase in subjects with arginase 1 deficiency (ARG1-D)

CONTACTS AND LOCATIONS:
Overall Officials: Cortney Caudill, Study Director — Aeglea BioTherapeutics, Inc.
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada